CLINICAL TRIAL: NCT04957316
Title: Effects of Removal of Endotoxin, Cytokines, and Uremic Toxins Using Blood Purification on Patients With Severe Septic Shock
Brief Title: Blood Purification in Patients With Septic Shock
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Collaborators: Baxter Healthcare Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202007010RIPD
Record Dates: First submitted 2021-06-23; First posted 2021-07-12 (Actual); Last update posted 2022-07-13 (Actual); Status verified 2022-07

CONDITIONS: Severe Septic Shock
MeSH Terms: conditions — Shock, Septic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): Conventional treatment of severe septic shock.
- Blood purification group (Experimental): Conventional treatment of severe septic shock and blood purification.
  Interventions: Device: Triple-effect blood purification filter

INTERVENTIONS:
Device: Triple-effect blood purification filter — Blood purification using the oXiris filter to remove endotoxin, cytokines, and uremic toxins.
  Arms: Blood purification group

SUMMARY:
In recent years, many studies have pointed out that bacterial toxin storm and cytokine storm are the main causes of patients with septic shock and multiple organ dysfunction. Endotoxins are the main mediators of gram-negative bacteria causing systemic inflammation and sepsis. Endotoxins can interact with Toll- Like receptor 4 (TLR4) binding and trigger cytokine storms. The triple-effect blood purification filter has been proven to remove endotoxins, cytokines and urinary toxins, and it has the opportunity to improve shock in patients with sepsis. We hypothesize that blood purification using the three-effect filter can shorten the duration and severity of shock in patients with severe septic shock and reduce the organ damage by removing endotoxin, cytokine and urinary toxins. The primary aim of this study is to investigate the effect of blood purification using the three-effect filter on shortening the duration of septic shock. Other exploratory variables include the reduction of severity of organ damage and other clinical outcomes and prognosis.

DETAILED DESCRIPTION:
In recent years, many studies have pointed out that bacterial toxin storm and cytokine storm are the main causes of patients with septic shock and multiple organ dysfunction. Endotoxins are the main mediators of gram-negative bacteria causing systemic inflammation and sepsis. Endotoxins can interact with Toll- Like receptor 4 (TLR4) binding and trigger cytokine storms. The triple-effect blood purification filter (oXiris) has been proven to remove endotoxins, cytokines and urinary toxins, and it has the opportunity to improve shock in patients with sepsis. We hypothesize that blood purification using the three-effect filter can shorten the duration and severity of shock in patients with severe septic shock and reduce the organ damage by removing endotoxin, cytokine and urinary toxins. The primary aim of this study is to investigate the effect of blood purification using the three-effect filter on shortening the duration of septic shock. Other exploratory variables include the reduction of severity of organ damage and other clinical outcomes and prognosis.

This multi-center, prospective, randomized controlled trial will enroll patient with septic shock. After the screening of eligibility and obtaining the signed informed consent, the enrolling patients will be randomly assigned to the following two groups: the control group and the blood purification group. In the control group, patients will receive the treatments for septic shock according to the Surviving Sepsis Campaign guidelines. If the primary care intensivist decides that continuous renal replacement therapy (CRRT) is indicated, the patient will receive CRRT with regular continuous veno-venous hemofiltration filter. In the blood purification group, patients will receive the treatments for septic shock according to the Surviving Sepsis Campaign guidelines. In addition, these patients will receive blood purification treatment with oXiris filter within two hours after enrollment. The blood purification treatment will be continued for up to 72 hours as needed, and a new oXiris filter will be replaced every 12 to 24 hours. If the primary care intensivist decides that continuous renal replacement therapy (CRRT) is indicated at 72h after blood purification, the patient will receive CRRT with regular continuous veno-venous hemofiltration filter.

The following information will be recorded: diagnosis of intensive care unit admission, past medical history, severity of illness, vital signs, blood pressure, infusion doses of vasopressors and inotropes, fluid balance, sequential organ failure assessment score, daily urine output, lactate, creatinine, and other regular laboratory data. Blood sample will be obtained for analysis of the levels of procalcitonin, cytokines (IL-6, IL-10, HMGB-1 and TNF-α), vascular endothelial cell injury biomarker, kidney injury biomarker and intestinal injury biomarkers.

The primary outcome is the difference of the duration of vasopressor between the two groups. The secondary is the proportion of reduction in vasoactive-inotropic score at 72h between the two groups. Other exploratory variables include the the proportion of reduction in vasoactive-inotropic score at other time points, the serum level of cytokines and organ injury biomarkers, and clinical outcomes between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* Critically ill patients with severe septic shock
* Intraabdominal infection, proved or highly suspected gram-negative bacteria infection
* Change of sequential organ failure assessment (SOFA) score is above or equal to 2
* Require norepinephrine infusion to maintain mean arterial pressure above 65 mm Hg
* Lactate level above 4 mmol/L
* SOFA score >= 9 or norepinephrine dose > 0.1 mcg/kg/min

Exclusion Criteria:

* Aged < 20
* SOFA score >=16
* Lactate level >=16
* High dose norepinephrine infusion (> 0.3 mcg/kg/min) more than 24 h after SOFA score was >=9
* High dose norepinephrine infusion (> 0.3 mcg/kg/min) more than 24 h after Lactate level was >=4
* White blood cell counts < 1000 cells/μL
* Platelet counts < 30 K/μL
* Allergy to heparin
* Receive continuous renal replacement therapy >8 hour before enrollment
* Receive other endotoxin removal filter
* Receive cardiopulmonary resuscitation within 4 weeks before enrollment
* Admitted to ICU for severe septic shock within 4 weeks before enrollment
* APACHE II score > 35 at enrollment

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2021-09-16 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Duration of vasopressors and inotropes infusion | up to 10 days
  Compare the duration of required infusion of vasopressors and inotropes between the two groups

SECONDARY OUTCOMES:
Proportion of reduction in vasoactive-inotropic score | 72 hours
  Compare the proportion of reduction in vasoactive-inotropic score (VIS) from enrollment to 72 hours after enrollment between the two groups. VIS = dopamine dose * 1 + dobutamine dose *1 + norepinephrine dose *100 + epinephrine dose * 100 + milrinone dose *10 + vasopressin dose x 10000. All above medication doses are calculated with the unit of mcg/kg/min.

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No